CLINICAL TRIAL: NCT05843877
Title: Pancreatic Head Resection or Total Pancreatectomy With Islet Autotransplantation (IAtx) in Patients With Periampullary Cancer and High Risk Profile for the Development of Postoperative Pancreatic Fistula (POPF)
Brief Title: Pancreatic Head Resection or Total Pancreatectomy With Islet Autotransplantation in Patients With Periampullary Cancer and High Risk Profile for the Development of Postoperative Pancreatic Fistula
Acronym: XandTX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUD-XandTX-079; 2023-507773-17-00 (EU CTIS Number)
Record Dates: First submitted 2023-02-27; First posted 2023-05-06 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Periampullary Cancer; Postoperative Pancreatic Fistula
MeSH Terms: interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Therapy (Experimental): Total pancreatectomy with autologous islet cell transplantation
  Interventions: Biological: Intraportal transplantation of isolated autologous pancreatic islets after total pancreatectomy
- Standard Therapy (Other): Pancreaticoduodenectomy (classic Whipple or pylorus-preserving)
  Interventions: Procedure: Pancreaticoduodenectomy (classic Whipple or pylorus-preserving)

INTERVENTIONS:
Biological: Intraportal transplantation of isolated autologous pancreatic islets after total pancreatectomy — Islet cells are isolated from patients healthy pancreatic tissue. Following total pancreatectomy, these autologous cells are injected into the portal vein, to implant in the liver and produce insulin.
  Arms: Experimental Therapy
Procedure: Pancreaticoduodenectomy (classic Whipple or pylorus-preserving) — As a standard procedure, the tumor-affected region of the pancreatic head with surrounding tissue and lymph nodes is removed during surgery. Reconstruction is performed by pancreaticojejunostomy.
  Arms: Standard Therapy

SUMMARY:
The primary objective of this clinical trial is to evaluate whether primary total pancreatectomy with simultaneous islet autotransplantation compared with pancreatic head resection (alone) can reduce perioperative morbidity and time to initiation of adjuvant therapy in patients with a high-risk constellation for pancreatic fistulas.

ELIGIBILITY:
Inclusion Criteria:

* suspected or confirmed periampullary carcinoma (tumor) and indication for PPPD (pylorus-preserving pancreaticoduodenectomy) or Whipple surgery
* high-risk profile for the development of a postoperative pancreatic fistula (POPF) after pancreatic head resection: soft pancreas and Pancreatic duct diameter < 3 mm (preoperative and intraoperative confirmation)
* written informed consent of the participant after successful Informed consent

Exclusion Criteria:

* patients on whom another procedure is to be performed simultaneously in addition to PPPD or Whipple surgery
* confirmed other primary tumor
* previous transplantation of an organ or tissue
* known infection with HIV (HIV antibodies)
* positive hepatitis C antibodies, positive hepatitis B surface antigens and hepatitis Bc antibodies
* insulin-treated diabetes mellitus
* history of hypersensitivity to any of the drugs used or their ingredients or to drugs with a similar chemical structure
* concurrent participation in another clinical trial (incl. within the last 4 weeks prior to inclusion).
* addiction or other medical conditions that do not allow the subject to understand the nature and not be able to appreciate the nature, scope and possible consequences of the trial
* pregnant or breastfeeding women
* women of childbearing age, except for women who meet the following criteria:

  1. Post-menopausal (12 months of natural amenorrhea or 6 months of amenorrhea with Serum FSH > 40 U/ml)
  2. Post-operative (6 weeks after bilateral ovariectomy with or without hysterectomy)
  3. Regular and correct use of a contraceptive method with an failure rate < 1% per year
  4. Sexual abstinence
  5. Vasectomy of the partner
* evidence that the patient is unlikely to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Duration between surgery and time "fit for adjuvant treatment" (postoperative day X) | From day of discharge until confirmed fitness for adjuvant treatment or 24 months, whichever came first
  Time (days) between surgery and the date of certified fitness to begin adjuvant therapy, confirmed by an oncology consult, starting at day of discharge, than assessed at POD 90, POD 180, POD 365, 24 months

SECONDARY OUTCOMES:
Comparison of actual start of adjuvant therapy in both arms | From POD 90 until actual start of therapy or 24 months whichever came first
  Postoperative day on which adjuvant therapy was started
Rate of peri-operative morbidity/mortality acc. to Clavien-Dindo classification | After enrolment of the patient until 24 months after intervention
  Rate of peri-operative morbidity/mortality will be assessed acc. to Clavien-Dindo classification
Rate of (serious) adverse events | After randomization of the patient until 24 months after intervention
  Rate of (serious) adverse events, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Version 5.0, 2017)
Patient reported outcomes: Quality of life EORTC QLQ C30 questionnaire | From date of screening until 24 months after intervention
  The QoL analyses will include QoL mean values, QoL response. EORTC QLQ C30 contains 30 questions28 questions regarding body fitness, daily routines, restrictions at work and hobby, appetite, fatigue, cough, breathlessness, pain, tiredness, and body conditions from (1) to (4); 1 (not a bit), 2 (little), 3 (moderate), 4 (much).
  2 questions regarding state of health and Quality of life with a horizontal rating from 1 to 7; 1 (very bad), 7 (excellent).; assessed at POD 90, POD 180, POD 365, and 24 months after surgery
Patient reported outcomes: Quality of life EORTC PAN26 questionnaire | From date of screening until 24 months after intervention
  The QoL analyses will include QoL mean values, QoL response. EORTC QLQ PAN26 contains 30 questions regarding pain, nutrition, body fitness, sexuality, from (1) to (4); 1 (not a bit), 2 (little), 3 (moderate), 4 (much).
  28 questions regarding body fitness, daily routines, restrictions at work and hobby, appetite, fatigue, cough, breathlessness, pain, tiredness, and body conditions from (1) to (4); 1 (not a bit), 2 (little), 3 (moderate), 4 (much); , assessed at POD 90, POD 180, POD 365, and 24 months after surgery
  2 questions regarding state of health and Quality of life with a horizontal rating from 1 to 7; 1 (very bad), 7 (excellent).
Comparison of metabolic outcome in both arms: continuous glucose monitoring (CGM) | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on continuous monitoring of glucose (CGM) in plasma (mmol/L) at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: glucagon | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on the hormone glucagon in plasma at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: glycohemoglobin HbA1c | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on glycohemoglobin (HbA1c in %) at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: C-peptide | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on serum C-peptide (nmol/L) as measure for functionality of pancreas at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: fructosamine | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on serum fructosamine (µmol/L) at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: insulin requirement | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on requirement of insulin (yes/no) at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: number of hypoglycemic events | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on number of hypoglycemic events (defined as value of blood glucose below 3.5 mmol/l) at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of metabolic outcome in both arms: severity of hypoglycemia | From date of screening until 24 months after intervention
  Metabolic outcome will be determined on severity of hypoglycemic events (decrease of blood glucose level) at every visit: Screening, POD 1, POD 3, day of discharge, POD 90, POD 180, POD 365 and 24 months after intervention
Comparison of long-term oncological course (24 months) in both arms: tumor markers | 24 months after intervention
  Within 24 months after intervention, oncological outcome is evaluated, as measured by tumor markers CA 19-9, CEA
Comparison of long-term oncological course (24 months) in both arms: recurrence | 24 months after intervention
  Within 24 months after intervention, oncological outcome is evaluated, as measured by recurrences of tumor shown in CT imaging
Comparison of long-term oncological course (24 months) in both arms: occurence of metastases | 24 months after intervention
  Within 24 months after intervention, oncological outcome is evaluated, as measured by metastases shown in CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Ludwig, Prof. Dr., Principal Investigator — Department of internal Medicine III; Marius Distler, Prof. Dr., Principal Investigator — Department of Visceral, Thoracic and Vascular Surgery
Locations (1):
- University Hospital Carl Gustav Carus Technische Universität Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hempel S, Kolbinger FR, Oehme F, Radulova-Mauersberger O, Schmid J, Schubert U, Schepp F, Bornstein S, Korn S, Trips E, Weitz J, Distler M, Ludwig B. Pancreatoduodenectomy versus total pancreatectomy and simultaneous intraportal islet autotransplantation for periampullary cancer at high-risk of postoperative pancreatic fistula (XANDTX-trial): Protocol of a randomized controlled pilot trial. PLoS One. 2025 Jul 28;20(7):e0327949. doi: 10.1371/journal.pone.0327949. eCollection 2025. PMID 40720532